CLINICAL TRIAL: NCT00927576
Title: PC-Based Cognitive Rehabilitation for TBI
Brief Title: PC-Based Cognitive Rehabilitation for Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B6119-R
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Traumatic Brain Injury
Keywords: cognitive training; neuroplasticity; cognitive impairment; recovery of function; memory; attention
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction | interventions — Trail Making Test

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control subjects: Control subjects = 237. These subjects underwent extensive testing with computerized neuropsychological tests including digit span testing, spatial span testing, simple reaction time testing, choice reaction time testing, finger tapping, verbal fluency, design fluency, verbal list learning, questionnaire completion, and the trail making test.
  Interventions: Behavioral: Digit span testing; Behavioral: Spatial span testing; Behavioral: Finger tapping; Behavioral: Simple reaction time; Behavioral: Choice reaction time; Behavioral: Verbal fluency; Behavioral: Verbal list learning; Behavioral: Trail making test; Behavioral: Design fluency; Behavioral: Questionnaire completion
- TBI patients: TBI patients N = 28. These patients underwent extensive testing with computerized neuropsychological tests including digit span testing, spatial span testing, simple reaction time testing, choice reaction time testing, finger tapping, verbal fluency, design fluency, verbal list learning, questionnaire completion, and the trail making test.
  Interventions: Behavioral: Digit span testing; Behavioral: Spatial span testing; Behavioral: Finger tapping; Behavioral: Simple reaction time; Behavioral: Choice reaction time; Behavioral: Verbal fluency; Behavioral: Verbal list learning; Behavioral: Trail making test; Behavioral: Design fluency; Behavioral: Questionnaire completion

INTERVENTIONS:
Behavioral: Digit span testing — Testing of short-term verbal memory with digit span
Behavioral: Spatial span testing — Testing of short-term visuospatial memory with spatial span.
Behavioral: Finger tapping — Testing motor speed with a finger tapping test.
Behavioral: Simple reaction time — Testing the time to respond to the appearance of a visual stimulus.
Behavioral: Choice reaction time — Testing the time needed to discriminate and respond to different visual stimuli.
Behavioral: Verbal fluency — Evaluating how many words are produced in 90s.
Behavioral: Verbal list learning — Evaluating short-term memory, learning, and memory interference in the recall of 12-word lists, presented three times. Evaluating long-term memory and recognition after a 20 min interval.
Behavioral: Trail making test — Evaluating visuomotor speed and executive function in Trail Making Tests, A and B. In the first, subjects connect successive numbers with the mouse. In the second, they connect numbers and letters in alternation.
Behavioral: Design fluency — Subjects create the maximal number of 4-line patterns in 90 s.
Behavioral: Questionnaire completion — Question completion time is measured on each question of the Post-Traumatic Stress Disorder check list (PCL) and on the cognitive failures questionnaire.

SUMMARY:
The investigators evaluated whether it was possible to improve the measurement of memory, attention, and executive function in patients who have suffered traumatic brain injury through the use of computer-based testing.

Note: the original design of the study was altered due to failure to recruit sufficient numbers of patients who were willing to undergo prolonged cognitive training.

DETAILED DESCRIPTION:
Here we describe a series of computer-based tests that were used to evaluate memory, attention, and executive function in large groups of control subjects and in patients with chronic mild and moderate/severe TBI. This extensive battery of neuropsychological tests (NPTs) and subjective rating scale measures were obtained at study entry from the TBI cohort. NPT and rating scale data were compared to those obtained from control subjects to characterize the cognitive deficits following mild, moderate and severe TBI. .

Normative data were obtained by regressing the influences of age, education, and computer use on scores to create normed z-scores on different NPTs,. We hypothesized that patient with TBI would show deficits on tests of memory, attention, and executive function relative to their predicted z-scores (based on the aforementioned regression functions) and that deficits would be more pronounced in patients with severe TBI than in patients with mild TBI.

ELIGIBILITY:
Inclusion Criteria:

Control subjects were required to meet the following inclusion criteria:

* (a) fluency in the English language
* (b) no current or prior history of bipolar disorder, mania, or schizophrenia
* (c) no current substance abuse
* (d) no concurrent history of neurologic disease known to affect cognitive functioning
* (e) on a stable dosage of any required medication
* (f) auditory functioning sufficient to understanding normal conversational speech and visual acuity normal or corrected to 20/40 or better

Exclusion criteria:

* History of TBI

Exclusion Criteria for TBI patients:

* TBI patients had to meet the same inclusion criteria as the controls with the exception that they were required to have a history of TBI. They also had to be in the chronic phase, i.e., 1-4 yrs post-injury.
* Exclusion criteria:

  * current substance abuse
  * current psychiatric diagnosis other than PTSD

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls subjects of various ages (approximately 230), and TBI patients (approximately 30).
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L. Woods, PhD, Principal Investigator — VA Northern California HCS

REFERENCES:
- [Background] Atkins Whitmer D, Woods DL. Analysis of the cost effectiveness of a suicide barrier on the Golden Gate Bridge. Crisis. 2013;34(2):98-106. doi: 10.1027/0227-5910/a000179. PMID 23261913
- [Background] Disbrow EA, Russo KA, Higginson CI, Yund EW, Ventura MI, Zhang L, Malhado-Chang N, Woods DL, Sigvardt KA. Efficacy of tailored computer-based neurorehabilitation for improvement of movement initiation in Parkinson's disease. Brain Res. 2012 May 3;1452:151-64. doi: 10.1016/j.brainres.2012.02.073. Epub 2012 Mar 9. PMID 22459048
- [Background] Whitaker KJ, Kang X, Herron TJ, Woods DL, Robertson LC, Alvarez BD. White matter microstructure throughout the brain correlates with visual imagery in grapheme-color synesthesia. Neuroimage. 2014 Apr 15;90:52-9. doi: 10.1016/j.neuroimage.2013.12.054. Epub 2014 Jan 7. PMID 24406309
- [Result] Woods DL, Herron TJ, Yund EW, Hink RF, Kishiyama MM, Reed B. Computerized analysis of error patterns in digit span recall. J Clin Exp Neuropsychol. 2011 Aug;33(7):721-34. doi: 10.1080/13803395.2010.550602. PMID 21957866
- [Result] Hubel KA, Reed B, Yund EW, Herron TJ, Woods DL. Computerized measures of finger tapping: effects of hand dominance, age, and sex. Percept Mot Skills. 2013 Jun;116(3):929-52. doi: 10.2466/25.29.PMS.116.3.929-952. PMID 24175464
- [Result] Hubel KA, Yund EW, Herron TJ, Woods DL. Computerized measures of finger tapping: reliability, malingering and traumatic brain injury. J Clin Exp Neuropsychol. 2013;35(7):745-58. doi: 10.1080/13803395.2013.824070. Epub 2013 Aug 15. PMID 23947782
- [Result] Woods DL, Kishiyamaa MM, Lund EW, Herron TJ, Edwards B, Poliva O, Hink RF, Reed B. Improving digit span assessment of short-term verbal memory. J Clin Exp Neuropsychol. 2011 Jan;33(1):101-11. doi: 10.1080/13803395.2010.493149. PMID 20680884

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Subjects | TBI Patients
Started | 237 | 28
Cognitive Testing | 237 | 28
Completed | 237 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Subjects: Control subjects = 230. Normal control subjects of various ages.
- TBI Patients: TBI patients N = 30. Mixed mild and severe TBI group, with most showing PTSD comorbidity.
- Total: Total of all reporting groups
Arm/Group | Control Subjects | TBI Patients | Total
Number analyzed (Participants) | 237 | 28 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 222 | 28 | 250
  >=65 years | 15 | 0 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (21.3) | 42.4 (10.3) | 41.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 1 | 108
  Male | 130 | 27 | 157
Region of Enrollment [Number; unit: participants] — Subjects from the San Francisco Bay Area
  participants
    United States | 237 | 28 | 265

OUTCOME MEASURES:

1. Primary Outcome: Performance in TBI Patients and Controls
Description: Subjects were assessed on a set of cognitive tests. Here we describe the results on the simple reaction time test in which subjects respond as rapidly as possible to the computer-controlled occurrence of a visual stimulus by pressing a mouse button. Two control groups were used. One large control group underwent a single test to provide data from subjects with a broad range of age and education. The other, smaller, control group underwent three tests at weekly intervals to evaluate the test-retest reliability of the measure.
Time Frame: Subjects were tested in a single 2-hr session.
Population: Data from two TBI patients were excluded due to suspected suboptimal effort.
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Simple Reaction Time Test: time to respond in ms to visual stimuli presented randomly to the left or right hemifield at varying stimulus onset asynchronies.
Arm/Group | Simple Reaction Time Test
Number analyzed (Participants) | 263
ms
  Control group 1, n=189 | 237.8 (27.8)
  Control group 2, n =48 | 231.5 (17.72)
  Mild TBI, n =22 | 228.0 (34.6)
  Severe TBI, n =4 | 280.0 (42.4)
Statistical Analysis 1: Comparison: Simple Reaction Time Test; The null hypotheses was that the severe TBI group would not differ from the control group in SRT latencies; Test type: Non-Inferiority or Equivalence — Power analysis of the results showed a 95% chance of finding a p<0.05 difference in 166 subjects and a 99% chance of finding a p <0.05 difference in 230 subjects in comparison of Group 1 controls and sTBI patients; p < 0.001, ANOVA; for repeated measures with effect sizes (omega squared); Difference in z-score, sTBI vs. controls = 2.04
Statistical Analysis 2: Comparison: Simple Reaction Time Test; The null hypothesis was that the mild TBI group would not differ in age-corrected z-score from that of a control subjects in the large control group; Test type: Non-Inferiority or Equivalence — Power analysis of controls (i.e., with z-score = 0) showed a 95% chance of detecting a p < 0.05 significance level for z-scores exceeding 0.54 in the mild TBI patient group; p = .50, ANOVA — The P-value reflects the likelihood of detection a difference of the magnitude observed; z-score difference between groups = -0.30

ADVERSE EVENTS:
Time Frame: Entire study duration (4 years).
Groups:
- Control Subjects: Control subjects = 237. No adverse events were observed.
- TBI Patients: TBI patients N = 28. No adverse events were observed
Arm/Group | Control Subjects | TBI Patients
Serious Adverse Events (participants affected / at risk) | 0/237 | 0/28
Other Adverse Events (participants affected / at risk) | 0/237 | 0/28

LIMITATIONS AND CAVEATS:
Relatively small TBI group limits strength of conclusions. Not all of the results have yet been fully analyzed and subjected to peer-review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes